CLINICAL TRIAL: NCT00321438
Title: Prospective, Observational Study of Subjects With CXCR4-Tropic or Non-Phenotypeable HIV to Assess Changes in Tropism Over Time
Brief Title: Observational Study of HIV-Infected Subjects With X4-Tropic or Non-Phenotypeable Virus
Status: Terminated | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: CCR104629
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: HIV Infection
Keywords: HIV-1; GW873140; CCR5 antagonist; experienced; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to measure viral tropism over time in subjects with X4-tropic or non-phenotypeable virus while receiving standard of care therapy. This is an observational study. No investigational treatment will be administered through this study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected.
* Screening viral load at least 5000copies/mL.
* X4-tropic only or non-phenotypeable virus at screening.
* Total prior antiretroviral experience of at least 3 months and documented resistance to at least one drug in each of the following classes: NRTI, NNRTI, and PI, stable antiretroviral regimen (or no antiretroviral treatment) for at least 4 weeks before screening.
* Able to receive a ritonavir-boosted protease inhibitor during treatment studies.
* Women of childbearing potential must use specific forms of contraception.

Exclusion criteria:

* R5-tropic only or R5/X4-tropic virus at screening, changes to antiretroviral therapy from 4 weeks prior to screening until Day 1 of observational study.
* Pregnant or breastfeeding women.
* Significant ECG abnormalities or significant history of active pancreatitis, hepatitis, opportunistic infections, cancer, or severe illness.
* Current use of certain medications may exclude participation in this study.
* Additional qualifying criteria and laboratory test requirements to be determined by study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (14):
- United States (14):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Key West, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hampton, Virginia